CLINICAL TRIAL: NCT01356329
Title: A Randomized, Controlled, Open Label Study of the Efficacy and Safety of the Low Molecular Weight Heparin (LMWH), LovenoxTM (Enoxaparin) Versus HeparinTM (Unfractionated Heparin) for Prevention of Venous Thromboembolism (VTE) in Gynecologic Oncology Patients
Brief Title: Efficacy and Safety of the LovenoxTM (Enoxaparin) Versus HeparinTM Gynecologic Oncology Patients
Acronym: Lovenox
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in enrolling patients
Sponsor: National Guard Health Affairs (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC08/118
Record Dates: First submitted 2011-03-19; First posted 2011-05-19 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Malignant Female Reproductive System Neoplasm
Keywords: Gynecologic malignancy ,major surgery
MeSH Terms: interventions — Enoxaparin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lovenox (Experimental): Group A : Low Molecular Weight Heparin (LMWH), LovenoxTM (Enoxaparin)
  Interventions: Drug: Enoxaparin, Heparin
- Heparin (Experimental): Group B:HeparinTM (Unfractionated Heparin)
  Interventions: Drug: Enoxaparin, Heparin

INTERVENTIONS:
Drug: Enoxaparin, Heparin — Patients who meet the Inclusion Criteria and signed an informed consent will be randomly assigned to 1 of the 2 treatment groups (the Enoxaparin (Group A) and Unfractionated Heparin (Group B)
  ). Subjects will be assigned consecutive study numbers according to a predetermined random code generated by the Biostatistician.

SUMMARY:
Prophylactic treatment will start from surgery until the patients are discharged from the hospital(18). Then each patient will have 2 follow up visit in gyne- oncology clinic. The first visit will be 2 weeks from discharge & the second visit will be 3 months after surgery. In each visit patient will be evaluated for any evidence of thrombo-embolic events clinically & radiologically if needed ( spiral CT, V/Q scan & lower limp Doppler ). Any side effect or adverse reaction will be reported & it will be evaluated if it is related to the drug used or not.

DETAILED DESCRIPTION:
This study is a phase IIIB, randomized, open label, non-comparative controlled trial, and prospectively enrolling 150 females to assess the efficacy and safety of the Enoxaparin (Group A) and Unfractionated Heparin (Group B) for Gynecologic Oncology Patients In the Kingdom of Saudi Arabia who required surgery or admission for the prevention of VTE.

Patients who meet the Inclusion Criteria and signed an informed consent will be randomly assigned to 1 of the 2 treatment groups (Group A or Group B). Subjects will be assigned consecutive study numbers according to a predetermined random code generated by the Biostatistician. The randomisation will be based on a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients aged 18 years or older were admitted with diagnosis of malignancy or suspension of malignancy and going for major surgery.
2. Patient with the following conditions:

   1. Any patient were admitted with diagnosis of Gynecologic malignancy & going for major surgery such as laparotomies & abdominal hysterectomy OR
   2. All staging laparotomies done for suspected ovarian malignancy by either ultrasound finding or tumor markers (raised CA 125) & found to be either borderline or benign ovarian tumor
3. Signed the Informed Consent Form

Exclusion Criteria:

1 Renal failure assessed by serum creatinine > 2.0mg/dL (180 mmol/L) 2. Patients on anticoagulant treatment in the previous 6 months 3. Bleeding disorders or platelet count < 80x109/L 4. Known hypersensitivity to unfractionated heparin or LMWHs 5. Pregnant women 6. Obese patients with body mass index ≥ 47

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Safety | 3 years
  Efficacy will be measured by measuring any thromboembolic events confirmed by objective testing such as spiral CT or V/Q scan and Doppler ultrasound as well as coagulation profile parameter, clinical sign and symptoms within 3 months post-operation.

SECONDARY OUTCOMES:
Safety | 3 years
  •To evaluate the Number of participants with Adverse Events and Serious Adverse Events of both treatment groups.
  Safety will include the following parameters for all patients who receive the study regimen:
  * Time to thromboembolic event
  * Total number of deaths from any cause
  * Proportion of patients with major bleeding
  * Site of thromboembolic event
  * Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Safi, MD, Principal Investigator — King Abdul Aziz Medical City for National Guard
Locations (1):
- King Abdul Aziz Medical City for National Guard Health Affairs, Riyadh, Saudi Arabia